CLINICAL TRIAL: NCT05342259
Title: Low Dose Caudal VS Dorsal Penile Nerve Block for Postoperative Analgesia After Circumcision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RAMY AHMED, Assistant Professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMASU MS 573/ 2021
Record Dates: First submitted 2022-03-08; First posted 2022-04-22 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- dorsal penile block patients (Active Comparator)
  Interventions: Procedure: Dorsal penile nerve block
- caudal block patients (Active Comparator)
  Interventions: Procedure: Caudal nerve block /neuroaxial
- combined block patients (Active Comparator)
  Interventions: Procedure: Combined caudal and dorsal penile nerve block

INTERVENTIONS:
Procedure: Caudal nerve block /neuroaxial — Technique of the caudal block The patient was placed in lateral decubitus position for blind caudal epidural block. A line was drawn to connect the bilateral posterior superior iliac crests and used as one side of an equilateral triangle; then the location of the sacral hiatus was approximated by palpating the sacral cornua as 2 bony prominences, the sacral hiatus was identified as a dimple in between. A needle was inserted at 45 degrees to the sacrum and redirected if the posterior surface of sacral bone was contacted.
  A subjective feeling of loss of resistance suggests piercing the sacral ligament.The "whoosh test," performed by auscultation at the thoracolumbar region with a stethoscope while injecting 2 mL of air, Palpating for subcutaneous bulging on rapid injection of 5 mL air or saline had a positive predictive value of 83% and a negative predictive value of 44%.
  Arms: caudal block patients
Procedure: Dorsal penile nerve block — Technique of Dorsal penile nerve block:
  Under aseptic technique and under ultrasound guidance. A 'hockey-stick' probe was used, covered by transparent sterile dressing. The probe was placed vertically over the pubic symphysis and the base of the penile shaft. With adjustment of the probe, a sagittal view of the penile shaft was produced. Scarpa's fascia was seen as a hyperechoic line superficial to the penile shaft. Under real-time guidance, the needle was inserted and advanced until its tip laid deep to Scarpa's fascia (i.e., within the subpubic space), where local anesthetic was deposited. The local anesthetic solution injected was 0.5% bupivacaine in a recommended volume. (2 ml up to 3 years and an additional 1 ml for each3 years up to maximum 6 ml).
  Arms: dorsal penile block patients
Procedure: Combined caudal and dorsal penile nerve block — Combined techniques of caudal and dorsal penile nerve block
  Arms: combined block patients

SUMMARY:
in order to eliminate fear and anxiety. Regional techniques are more effective than systemic opioids, non steroidal anti-inflammatory drugs, and acetaminophen for postoperative analgesia in circumcision, The most preferred techniques are dorsal penile nerve block and caudal block.

Objective: To investigate the effectiveness of post operative analgesia and complications among dorsal penile nerve block, caudal block and the combination of both.

Patients and Methods: Our study was carried out to compare the effectiveness, duration of post-operative analgesia, and the complications among dorsal penile nerve block (DPNB), caudal nerve block (CNB) and the combination of both. This study will carrey out on 81 male patients, aged from 3-12 years old & undergoing circumcision. The patients were divided into 3 groups, each is composed of 27 patients; group 1 including DPNB patients, group 2 including CNB patients and group 3 for combined block. This study compared between the three groups regarding the intra-operative vital data (HR,BP), post-operative VAS scores and the complications (nausea, vomiting, urinary retention, itching, constipation & CNS depression).

DETAILED DESCRIPTION:
Cases were subdivided into three groups: Group 1: included dorsal penile block patients. Group 2: included caudal block patients. Group 3: included combined block patients.

Circumcision was performed under general anesthesia and dorsal slit technique was used.

Study procedure:

General anesthesia was induced and maintained by inhalation of sevoflurane in oxygen mixed with air gas flow. A 22-G intravenous (i.v.) cannula was placed after induction. Spontaneous respiration was maintained via a selected laryngeal mask airway, and the inhaled sevoflurane was modified and maintained as 0.8 to 1.0MAC.

Block techniques:

Technique of the caudal block The patient was placed in lateral decubitus position for blind caudal epidural block. A line was drawn to connect the bilateral posterior superior iliac crests and used as one side of an equilateral triangle; then the location of the sacral hiatus was approximated by palpating the sacral cornua as 2 bony prominences, the sacral hiatus was identified as a dimple in between. A needle was inserted at 45 degrees to the sacrum and redirected if the posterior surface of sacral bone was contacted.

A subjective feeling of loss of resistance suggests piercing the SCL but was associated with a miss rate up to 26% even in experienced hands. The "whoosh test," performed by auscultation at the thoracolumbar region with a stethoscope while injecting 2 mL of air, had a sensitivity of 80% and a specificity of 60% in adults. Palpating for subcutaneous bulging on rapid injection of 5 mL air or saline had a positive predictive value of 83% and a negative predictive value of 44%. The inaccuracy of using blind technique for caudal epidural injection in adults, even confirmed by various tests, is clearly evident.

Drugs and doses used: 0.5 ml/kg of 0.25% Bupivacaine (diluted by saline solution 0.9).

Technique of Dorsal penile nerve block:

Under aseptic technique and under ultrasound guidance. A 'hockey-stick' probe was used, covered by transparent sterile dressing. The probe was placed vertically over the pubic symphysis and the base of the penile shaft. With adjustment of the probe, a sagittal view of the penile shaft was produced. Scarpa's fascia was seen as a hyperechoic line superficial to the penile shaft. Under real-time guidance, the needle was inserted and advanced until its tip laid deep to Scarpa's fascia (i.e., within the subpubic space), where local anesthetic was deposited. The local anesthetic solution injected was 0.5% bupivacaine in a recommended volume. (2 ml up to 3 years and an additional 1 ml for each3 years up to maximum 6 ml). Combined block:

The caudal block was performed then the patient was placed in supine position and the DPNB was done .

ELIGIBILITY:
Inclusion Criteria:

* Age: 3-12 years.
* ASA I & II.

Exclusion Criteria:

* Patient's refusal.
* Contraindications to regional blocks as bleeding disorders and skin infections.
* Drug hypersensitivity.
* Failure of achieving block.

Ages: 3 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 81 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
pain scoring using the Wong Baker scale | 1st hour postoperatively
  scale at 1st hour post operative, that shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable". Based on the faces and written descriptions, the patient chooses the face that best describes their level of pain.
pain scoring using the Wong Baker scale | 3rd hour postoperatively
  scale at 3rd hour post operative, that shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable". Based on the faces and written descriptions, the patient chooses the face that best describes their level of pain.
pain scoring using the Wong Baker scale | 24th hour postoperatively
  scale at 24th hour post operative, that shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable". Based on the faces and written descriptions, the patient chooses the face that best describes their level of pain.

SECONDARY OUTCOMES:
: intra-operative heart rate (beats/ minuts). | scale at 1st hour post operative
: intra-operative heart rate (beats/ minuts). | scale at 3rd hour post operative
: intra-operative heart rate (beats/ minuts). | scale at 24th hour post operative
intra-operative mean arterial blood pressure (mmhg) | intraoperatively
complications | one day after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No